CLINICAL TRIAL: NCT01644500
Title: The Efficacy and Safety of Once-Weekly, Subcutaneous Dulaglutide Monotherapy Compared to Glimepiride in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study Comparing the Effects and Safety of Dulaglutide With Glimepiride in Type 2 Diabetes Mellitus
Acronym: AWARD-CHN1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11991; H9X-JE-GBCG (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; glimepiride; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1.5 mg Dulaglutide (Experimental): 1.5 milligrams (mg) dulaglutide administered as one subcutaneous (SC) injection once-weekly plus one to three capsules of placebo each day for blinding purposes for up to 26 weeks.
  Interventions: Drug: Dulaglutide; Drug: Placebo as Capsules
- 0.75 mg Dulaglutide (Experimental): 0.75 mg dulaglutide administered as one SC injection once-weekly plus one to three capsules of placebo each day for blinding purposes for up to 26 weeks.
  Interventions: Drug: Dulaglutide; Drug: Placebo as Capsules
- Glimepiride (Active Comparator): 1 to 3 mg per day (mg/day) glimepiride administered orally as one to three capsules per day plus one SC injection of placebo once-weekly for blinding purposes for up to 26 weeks.
  Interventions: Drug: Glimepiride; Drug: Placebo as SC Injection

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 0.75 mg Dulaglutide; 1.5 mg Dulaglutide
Drug: Glimepiride — Administered orally
  Arms: Glimepiride
Drug: Placebo as Capsules — Placebo for glimepiride is administered orally as one to three capsules daily.
  Arms: 0.75 mg Dulaglutide; 1.5 mg Dulaglutide
Drug: Placebo as SC Injection — Placebo for dulaglutide is administered as one SC injection.
  Arms: Glimepiride

SUMMARY:
The purpose of this study is to examine if once-weekly dulaglutide is efficient and safe compared to glimepiride in participants with type 2 diabetes mellitus who have inadequate glycemic control with oral antihyperglycemic medication (OAM) or are OAM-naïve.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* OAM-naïve or have been taking OAM monotherapy for at least 3 months
* Glycosylated Hemoglobin (HbA1c) value of ≥7.0% to ≤10.5% for OAM-naïve participants or ≥6.5% to ≤10.0% for participants taking OAM monotherapy
* Adult men or adult non-pregnant, non-breastfeeding women
* Stable weight (±5%) ≥3 months prior to screening
* Body mass index (BMI) of ≥19.0 to ≤35.0 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have previously been treated with a glucagon-like peptide-1 (GLP-1) receptor agonist, GLP-1 analog, or any other incretin mimetic during the 3 months before screening
* Are currently taking dipeptidylpeptidase-IV (DPP-IV) inhibitor and thiazolidinediones (TZD) during the 3 months before screening
* Have gastric emptying abnormality
* Have cardiac disorder defined as unstable angina, myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, heart failure, arrhythmia, transient ischemic attack, or stroke
* Have poorly controlled hypertension (systolic blood pressure above 160 millimeters of mercury [mmHg] or diastolic blood pressure above 95 mmHg)
* Have impaired liver function
* Have impaired kidney function
* Have history of chronic pancreatitis or acute pancreatitis
* Have a serum calcitonin ≥20 picogram/milliliter (pg/mL)
* Have a personal or family history of medullary C-cell hyperplasia, focal hyperplasia, carcinoma or multiple endocrine neoplasia type 2 (MEN 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (30):
- China (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guiyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huai'an
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanning
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Qingdao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shijiazhuang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuxi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xiamen
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gangwon-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeju Special Self-Governing Pr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yong Kung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Kuang J, Zhu J, Liu S, Li Q. Efficacy and Safety of Once-Weekly Dulaglutide in Elderly Chinese Patients with Type 2 Diabetes: A Post Hoc Analysis of AWARD-CHN Studies. Diabetes Ther. 2020 Oct;11(10):2329-2339. doi: 10.1007/s13300-020-00910-1. Epub 2020 Aug 28. PMID 32857293
- [Derived] Guo L, Zhang B, Hou J, Zhou Z. Evaluation of Characteristics of Gastrointestinal Adverse Events with Once-Weekly Dulaglutide Treatment in Chinese Patients with Type 2 Diabetes: A Post Hoc Pooled Analysis of Two Randomized Trials. Diabetes Ther. 2020 Aug;11(8):1821-1833. doi: 10.1007/s13300-020-00869-z. Epub 2020 Jul 4. PMID 32621083
- [Derived] Yu M, Yuan GY, Zhang B, Wu HY, Lv XF. Efficacy and Safety of Dulaglutide by Baseline HbA1c in Chinese Patients with Type 2 Diabetes: A Post Hoc Analysis. Diabetes Ther. 2020 May;11(5):1147-1159. doi: 10.1007/s13300-020-00804-2. Epub 2020 Apr 10. PMID 32277401
- [Derived] Li YM, Zhang LH, Li XJ, Zhang B, Hou JN, Tong NW. Efficacy and Safety of Dulaglutide Monotherapy Compared to Glimepiride in Oral Antihyperglycemic Medication-Naive Chinese patients with Type 2 Diabetes: A Post Hoc Analysis of AWARD-CHN1. Diabetes Ther. 2020 May;11(5):1077-1090. doi: 10.1007/s13300-020-00799-w. Epub 2020 Mar 26. PMID 32219675
- [Derived] Li H, Xu X, Wang J, Kong X, Chen M, Jing T, Zhang Z, Yin G, Liu X, Hu Y, Ye L, Su X, Ma J. A Randomized Study to Compare the Effects of Once-Weekly Dulaglutide Injection and Once-Daily Glimepiride on Glucose Fluctuation of Type 2 Diabetes Mellitus Patients: A 26-Week Follow-Up. J Diabetes Res. 2019 Apr 30;2019:6423987. doi: 10.1155/2019/6423987. eCollection 2019. PMID 31183384

RESULTS

PARTICIPANT FLOW:
Groups:
- Glimepiride: 1 to 3 mg/day glimepiride administered orally as one to three capsules per day plus one SC injection of placebo once-weekly for blinding purposes for up to 26 weeks.
Period: Overall Study
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Started | 244 | 248 | 245
Received at Least One Dose of Study Drug | 244 | 248 | 243
Modified Intent-to-treat Population | 239 | 239 | 242
Completed | 222 | 224 | 230
Not Completed | 22 | 24 | 15
Not completed — Adverse Event | 6 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 8 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 12 | 12
Not completed — Physician Decision | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is reported for the modified intent-to-treat population, who are all randomized participants with a baseline glycosylated hemoglobin (HbA1c) measurement, with at least 1 post-baseline HbA1c measurement, and who received at least one dose of study drug.
Groups:
- 1.5 mg Dulaglutide: 1.5 mg dulaglutide administered as one SC injection once-weekly plus one to three capsules of placebo each day for blinding purposes for up to 26 weeks.
- Total: Total of all reporting groups
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride | Total
Number analyzed (Participants) | 239 | 239 | 242 | 720
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.69 (10.754) | 53.79 (10.093) | 51.97 (10.052) | 52.81 (10.317)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 112 | 112 | 329
  Male | 134 | 127 | 130 | 391
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 239 | 239 | 242 | 720
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 29 | 28 | 29 | 86
  China | 184 | 186 | 186 | 556
  South Korea | 26 | 25 | 27 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at 26 Weeks
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline HbA1c as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, and had at least one post-baseline HbA1c measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
percentage of HbA1c | -1.48 (0.069) | -1.22 (0.069) | -0.92 (0.069)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.58, 95% CI 2-sided [-0.76 to -0.39]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.50 to -0.13]

2. Secondary Outcome: Percentage of Participants Attaining HbA1c of <7% or ≤6.5% at 26 Weeks
Description: Percentages of participants who achieved HbA1c levels of <7% or ≤6.5% were analyzed using a logistic regression model, controlling for treatment, pre-treatment, baseline HbA1c and country.
Time Frame: 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, and had at least one post-baseline HbA1c measurement. Last observation carried forward (LOCF) methodology was used to impute missing post-baseline values.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
percentage of participants
  HbA1c ≤6.5% | 59.4 | 47.7 | 41.3
  HbA1c <7.0% | 74.1 | 63.6 | 57.4
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Fisher Exact — Treatment comparison for HbA1c ≤6.5%; Odds Ratio (OR) = 2.7, 05% CI 2-sided [1.8 to 4.1]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Fisher Exact — Treatment comparison for HbA1c ≤6.5%; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.0 to 2.3]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Fisher Exact — Treatment comparison for HbA1c <7.0%; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.8 to 4.5]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.192, Fisher Exact — Treatment comparison for HbA1c <7.0%; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.1 to 2.5]

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at 26 Weeks
Description: FBG is a test to determine how much glucose (sugar) is in a blood sample after an overnight fast. FBG was measured by a central laboratory. LS means were calculated using MMRM analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline FBG as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
millimoles per liter (mmol/L) | -2.71 (0.135) | -2.26 (0.137) | -1.89 (0.136)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.83, 95% CI 2-sided [-1.15 to -0.51]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.70 to -0.05]

4. Secondary Outcome: Change From Baseline in 7-point Self-monitored Blood Glucose (SMBG) Profiles at 26 Weeks
Description: Change from baseline in mean daily blood glucose (BG) values were measured with a 7-point SMBG profile. Participants recorded their 7-point SMBG profiles on 2 separate, non-consecutive days during the 2-week period immediately before randomization, Week 8, Week 16, and Week 26 (or the Early Discontinuation Visit). The 7-point SMBG profile consisted of pre-prandial BG measures before the morning (fasting), midday, and evening meals; BG measures 2 hours after the start (post-prandial) of the morning, midday, and evening meals; and BG measures at bedtime. Mean at 26 weeks was assessed in all treatment groups. LS means were calculated using MMRM analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline body weight as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
mmol/L
  Morning (fasting) | -2.47 (0.092) | -1.91 (0.092) | -1.80 (0.091)
  Morning (2 hours post-prandial) meal | -4.56 (0.180) | -3.75 (0.181) | -3.20 (0.179)
  Midday (pre-prandial) meal | -3.09 (0.151) | -2.43 (0.151) | -2.37 (0.150)
  Midday (2 hours post-prandial) meal | -4.15 (0.174) | -3.40 (0.174) | -2.58 (0.173)
  Evening (pre-prandial) meal | -2.36 (0.135) | -1.77 (0.136) | -1.69 (0.134)
  Evening (2 hours post-prandial) meal | -3.63 (0.164) | -2.80 (0.165) | -2.35 (0.164)
  Bedtime | -3.22 (0.152) | -2.69 (0.152) | -2.03 (0.150)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for morning (fasting); Mean Difference (Net) = -0.67, 95% CI 2-sided [-0.89 to -0.45]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.304, Mixed Models Analysis — Treatment comparison for morning (fasting); Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.34 to 0.11]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for morning (2 hours post-prandial) meal; Mean Difference (Net) = -1.36, 95% CI 2-sided [-1.80 to -0.92]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — Treatment comparison for morning (2 hours post-prandial) meal; Mean Difference (Net) = -0.55, 95% CI 2-sided [-0.99 to -0.11]
Statistical Analysis 5: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for midday (pre-prandial) meal; Mean Difference (Net) = -0.73, 95% CI 2-sided [-1.10 to -0.36]
Statistical Analysis 6: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.740, Mixed Models Analysis — Treatment comparison for midday (pre-prandial) meal; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.43 to 0.31]
Statistical Analysis 7: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of midday (2 hours post-prandial) meal; Mean Difference (Net) = -1.56, 95% CI 2-sided [-1.99 to -1.13]
Statistical Analysis 8: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of midday (2 hours post-prandial) meal; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.24 to -0.39]
Statistical Analysis 9: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for evening (pre-prandial) meal; Mean Difference (Net) = -0.67, 95% CI 2-sided [-1.00 to -0.34]
Statistical Analysis 10: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.638, Mixed Models Analysis — Treatment comparison for evening (pre-prandial) meal; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.41 to 0.25]
Statistical Analysis 11: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for evening (2 hours post-prandial) meal; Mean Difference (Net) = -1.27, 95% CI 2-sided [-1.68 to -0.87]
Statistical Analysis 12: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — Treatment comparison for evening (2 hours post-prandial) meal; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.85 to -0.04]
Statistical Analysis 13: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for bedtime; Mean Difference (Net) = -1.19, 95% CI 2-sided [-1.56 to -0.82]
Statistical Analysis 14: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for bedtime; Mean Difference (Net) = -0.66, 95% CI 2-sided [-1.03 to -0.29]

5. Secondary Outcome: Rate of Hypoglycemic Episodes
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or documented BG concentrations of ≤70 milligrams per deciliter (mg/dL) (≤3.9 mmol/L). A severe hypoglycemic episode was defined as any hypoglycemic event for which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Nocturnal hypoglycemia is defined as any hypoglycemic event that occurs between bedtime and waking. Log mean rates of total hypoglycemia (per 30 days per participant) are presented and were calculated from negative binomial regression model. The model included country/region, prior medication group, treatment, visit, and treatment-by-visit interaction. The logarithm of days between visits was adjusted as an offset to account for possible unequal duration between visits and between participants.
Time Frame: Baseline through 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, and had evaluable hypoglycemic data.
Measure: Mean (Standard Deviation); unit: episodes/participant/30 days
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 244 | 247 | 243
episodes/participant/30 days
  All Hypoglycemic Episodes | 0.01 (0.053) | 0.01 (0.041) | 0.09 (0.581)
  Severe Hypoglycemic Episodes | NA (NA) — Data not available because no severe hypoglycemic episodes occurred. | NA (NA) — Data not available because no severe hypoglycemic episodes occurred. | NA (NA) — Data not available because no severe hypoglycemic episodes occurred.
  Nocturnal Hypoglycemic Episodes | 0.00 (0.011) | 0.00 (0.010) | 0.01 (0.057)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Negative binomial regression model — Treatment comparison for all hypoglycemic episodes
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Negative binomial regression model — Treatment comparison for all hypoglycemic episodes
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.008, Negative binomial regression model — Treatment comparison for nocturnal hypoglycemic episodes. Nocturnal hypoglycemic episodes are rounded off to 2 decimal places
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.006, Negative binomial regression model — [p-value comment as in outcome 5, analysis 3]

6. Secondary Outcome: Number of Participants With Self-Reported Hypoglycemic Episodes
Description: The overall number of participants with self-reported hypoglycemic episodes is presented.
Time Frame: Baseline through 26 Weeks
Population: All participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 244 | 248 | 243
participants | 14 | 9 | 38
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Fisher Exact

7. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment 2 Steady-state Beta (β) - Cell Function (HOMA2-%B) at 26 Weeks
Description: Change from baseline in HOMA2-%B was assessed by using the homeostasis model assessment (HOMA) to quantify β-cell function. HOMA2-%B is a computer model that uses FBG, insulin, and C-peptide concentrations to estimate steady state β-cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. LS means were calculated using an analysis of covariance (ANCOVA) model with country, baseline, pre-treatment, and treatment as fixed effects.
Time Frame: Baseline, up to 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, and had at least one post-baseline HbA1c measurement. LOCF methodology was used to impute missing post-baseline values.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%B
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
percentage of HOMA2-%B
  Insulin-based HOMA-2%B | 47.40 (2.624) | 37.92 (2.664) | 30.00 (2.591)
  C-peptide HOMA-2%B | 41.02 (1.945) | 34.57 (1.974) | 24.58 (1.964)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Insulin HOMA2-%B; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 17.41, 95% CI 2-sided [11.27 to 23.55]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Insulin HOMA2%B; Test type: Superiority or Other; p = 0.012, ANCOVA; Mean Difference (Net) = 7.92, 95% CI 2-sided [1.78 to 14.06]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Glimepiride; C-Peptide-Based HOMA2-%B; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 16.44, 95% CI 2-sided [11.81 to 21.06]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Glimepiride; C-Peptide-Based HOMA2-%B; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 9.99, 95% CI 2-sided [5.36 to 14.62]

8. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment 2 Insulin Sensitivity - Cell Function (HOMA2-%S) at 26 Weeks
Description: Change from baseline in HOMA2-%S was assessed by using the HOMA to quantify insulin sensitivity. HOMA2-%S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state insulin sensitivity (%S) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. LS means were calculated using an ANCOVA model with country, baseline, pre-treatment, and treatment as fixed effects.
Time Frame: Baseline, up to 26 Weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%S
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
percentage of HOMA2-%S
  Insulin-Based HOMA2-%S | -6.85 (2.636) | -10.33 (2.662) | -7.19 (2.602)
  C-Peptide-Based HOMA2-%S | -6.44 (2.056) | -11.84 (2.082) | -5.05 (2.074)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Insulin-Based HOMA2%S; Test type: Superiority or Other; p = 0.913, ANCOVA; Mean Difference (Net) = 0.34, 95% CI 2-sided [-5.83 to 6.51]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Insulin-Based HOMA2%S; Test type: Superiority or Other; p = 0.318, ANCOVA; Mean Difference (Net) = -3.14, 95% CI 2-sided [-9.30 to 3.03]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Glimepiride; C-Peptide-Based HOMA2-%S; Test type: Superiority; p = 0.576, ANCOVA; Mean Difference (Net) = -1.39, 95% CI 2-sided [-6.27 to 3.49]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Glimepiride; C-Peptide-Based HOMA2-%S; Test type: Superiority; p = 0.007, ANCOVA; Mean Difference (Net) = -6.79, 95% CI 2-sided [-11.68 to -1.89]

9. Secondary Outcome: Change From Baseline in Pancreatic Enzymes at 26 Weeks
Description: Amylase (total and pancreas-derived) and lipase concentrations were measured.
Time Frame: Baseline, 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, had at least one post-baseline HbA1c measurement and had evaluable pancreatic enzyme data.
Measure: Mean (Standard Deviation); unit: units per liter (u/L)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
units per liter (u/L)
  Total amylase | 9.29 (16.237) | 7.04 (13.128) | 3.79 (12.538)
  Pancreas-derived amylase | 6.19 (12.824) | 4.92 (8.123) | 2.64 (8.218)
  Lipase | 10.62 (30.086) | 9.28 (22.651) | 2.38 (22.717)

10. Secondary Outcome: Change From Baseline in Serum Calcitonin at 26 Weeks
Time Frame: Baseline, 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, had at least one post-baseline HbA1c measurement, and had evaluable serum calcitonin data.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
picomoles per liter (pmol/L) | -0.01 (0.318) | -0.02 (0.298) | 0.02 (1.193)

11. Secondary Outcome: Change From Baseline in Sitting Blood Pressure at 26 Weeks
Description: Sitting systolic blood pressure (SBP) and sitting diastolic blood pressure (DBP) were measured. LS means were calculated using MMRM analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline blood pressure as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: All participants who were randomized, received at least one dose of study drug, and had evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 222 | 224 | 231
millimeters of mercury (mmHg)
  SBP | -2.07 (0.815) | -1.88 (0.813) | -0.66 (0.804)
  DBP | -0.10 (0.535) | -0.11 (0.534) | 0.15 (0.526)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.180, Mixed Models Analysis — Treatment comparison for SBP
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.245, Mixed Models Analysis — Treatment comparison for SBP
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.717, Mixed Models Analysis — Treatment comparison for DBP
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.619, Mixed Models Analysis — Treatment comparison for DBP

12. Secondary Outcome: Change From Baseline in Sitting Pulse Rate at 26 Weeks
Description: LS means were calculated using MMRM analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline pulse rate as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: All participants who were randomized, received at least one dose of study drug, and had evaluable pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 222 | 224 | 231
beats per minute (bpm) | 3.07 (0.581) | 1.24 (0.581) | -0.34 (0.572)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis

13. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters, Fridericia Corrected QT (QTcF) Interval and P-R Wave (PR) Interval at 26 Weeks
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTcF = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and R-R wave (RR), which is the interval between two R waves. PR is the interval between the P wave and the ventricular depolarization wave (QRS) complex.
Time Frame: Baseline, 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, had at least one post-baseline HbA1c measurement, and had evaluable ECG data.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
milliseconds (msec)
  QT interval | -6.18 (21.469) | -2.06 (19.549) | 1.21 (23.021)
  PR interval | 3.73 (13.411) | 3.29 (11.236) | -0.23 (10.184)

14. Secondary Outcome: Change From Baseline in Heart Rate From ECG at 26 Weeks
Time Frame: Baseline, 26 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
bpm | 3.99 (8.459) | 1.90 (8.046) | 0.44 (9.275)

15. Secondary Outcome: Change From Baseline in Body Weight at 26 Weeks
Description: LS means were calculated using MMRM analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline body weight as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: All participants who were randomized, received at least one dose of study drug, and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 222 | 224 | 231
kilogram (kg) | -1.46 (0.192) | -0.77 (0.192) | 0.89 (0.190)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

16. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at 26 Weeks
Description: BMI is an estimate of body fat based on body weight divided by height squared. LS means were calculated using MMRM analysis adjusting for treatment, country, pre-study therapy stratum, visit, and treatment-by-visit as fixed effects; baseline body weight as covariate; and participant as a random effect.
Time Frame: Baseline, 26 Weeks
Population: All participants who were randomized, received at least one dose of study drug, and had evaluable BMI data.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 222 | 223 | 231
kilograms per meter squared (kg/m^2) | -0.55 (0.070) | -0.29 (0.070) | 0.32 (0.069)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Glimepiride; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

17. Secondary Outcome: Percentage of Participants Developing Antibodies to Dulaglutide
Description: Dulaglutide anti-drug antibodies (ADA) were assessed at baseline and 26 weeks. A participant was considered to have treatment-emergent dulaglutide ADA if the participant had at least 1 titer that was treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline through 26 Weeks
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, had at least one post-baseline HbA1c measurement, and had evaluable ADA data.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
percentage of participants | 17 | 8 | 4

18. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events
Description: Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular AEs that were adjudicated included myocardial infarction; hospitalization for unstable angina; hospitalization for heart failure; coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention); and cerebrovascular events, including cerebrovascular accident (stroke) and transient ischemic attack. A summary of serious and other non-serious AEs regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
number of participants | 0 | 1 | 0

19. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis
Description: The number of adjudicated (by an independent committee of expert physicians) pancreatic events is summarized at 26 weeks. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
participants | 7 | 5 | 1

20. Secondary Outcome: European Quality of Life Questionnaire-5 Dimensions (EQ-5D) Health State Score Responses at 26 Weeks
Description: The EQ-5D questionnaire is a widely used, generic questionnaire that assesses 5 dimensions associated with quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 3 possible levels of response: no problem, some problem, and extreme problem. Additional categories of response include ambiguous and missing. The number of participants per each of the 5 response categories is summarized for each of the 5 dimensions.
Time Frame: Week 26
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, had at least one post-baseline HbA1c measurement, and had evaluable EQ-5D data.
Measure: Number; unit: participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 239 | 239 | 242
participants
  Mobility - no problem | 217 | 218 | 224
  Mobility - some problem | 4 | 3 | 6
  Mobility - extreme problem | 0 | 0 | 0
  Mobility - ambiguous | 0 | 0 | 0
  Mobility - missing | 1 | 3 | 1
  Self-care - no problem | 221 | 220 | 228
  Self-care - some problem | 0 | 1 | 2
  Self-care - extreme problem | 0 | 0 | 0
  Self-care - ambiguous | 0 | 0 | 0
  Self-care - missing | 1 | 3 | 1
  Usual activities - no problems | 221 | 219 | 228
  Usual activities - some problems | 0 | 2 | 2
  Usual activities - extreme problems | 0 | 0 | 0
  Usual activities - ambiguous | 0 | 0 | 0
  Usual activities - missing | 1 | 3 | 1
  Pain/Discomfort - no problems | 198 | 192 | 200
  Pain/Discomfort - some problems | 23 | 28 | 29
  Pain/Discomfort - extreme problems | 0 | 0 | 0
  Pain/Discomfort - ambiguous | 0 | 0 | 0
  Pain/Discomfort - missing | 1 | 3 | 1
  Anxiety/Depression - no problems | 208 | 214 | 213
  Anxiety/Depression - some problems | 13 | 7 | 17
  Anxiety/Depression - extreme problems | 0 | 0 | 0
  Anxiety/Depression - ambiguous | 0 | 0 | 0
  Anxiety/Depression - missing | 1 | 3 | 1

21. Secondary Outcome: Visual Analog Scale (VAS) Score at 26 Weeks
Description: The EQ-5D questionnaire is a widely used, generic questionnaire that assesses health-related quality of life and consists of a 100-milliliter (mm) visual analog scale (VAS) on which the participant rated their perceived health state on that day from 0-mm (worst imaginable health state) to 100-mm (best imaginable health state).
Time Frame: Week 26
Population: Participants who had been randomized, received at least one dose of study drug, had a baseline HbA1c measurement, had at least one post-baseline HbA1c measurement, and had evaluable VAS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Number analyzed (Participants) | 234 | 230 | 237
units on a scale | 85.72 (9.723) | 86.17 (10.744) | 85.96 (10.938)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Glimepiride
Serious Adverse Events (participants affected / at risk) | 6/244 | 4/248 | 3/243
Other Adverse Events (participants affected / at risk) | 165/244 | 141/248 | 137/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=244) | 0.75 mg Dulaglutide (N=248) | Glimepiride (N=243)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract diabetic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=244) | 0.75 mg Dulaglutide (N=248) | Glimepiride (N=243)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Type iia hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eyelids pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Normal tension glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 5 (9) | 2 (2) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 16 (20) | 6 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 6 (7) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 7 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 42 (59) | 18 (20) | 7 (10)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 2 (5) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 2 (3) | 2 (5) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (7) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (6) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 25 (26) | 13 (14) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 19 (20) | 4 (5) | 1 (1)
Asthenia (General disorders) | 1 (1) | 3 (3) | 5 (6)
Chest discomfort (General disorders) | 4 (4) | 2 (2) | 2 (2)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (2) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 16 (21) | 13 (15) | 13 (13)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rabies (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 8 (8) | 11 (11)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 6 (6)
Vaginal infection (Infections and infestations) | 0/109 (0) | 1/114 (1) | 0/112 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (4) | 1 (1) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Albumin urine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 9 (16) | 6 (6) | 1 (1)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood creatinine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram st-t change (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Gastric ph decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Haematology test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 15 (19) | 14 (14) | 6 (6)
Lipids increased (Investigations) | 2 (2) | 4 (4) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein urine (Investigations) | 1 (1) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 3 (3)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Sinus rhythm (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Urine leukocyte esterase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine protein/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 2 (2) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 13 (13) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 9 (9) | 9 (9) | 10 (10)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 27 (27) | 30 (30) | 41 (41)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (5)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 4 (5)
Headache (Nervous system disorders) | 5 (8) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/135 (1) | 0/134 (0) | 0/131 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/109 (0) | 2/114 (5) | 0/112 (0)
Menorrhagia (Reproductive system and breast disorders) | 1/109 (1) | 0/114 (0) | 0/112 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/109 (0) | 1/114 (1) | 0/112 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne varioliformis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Yellow skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Papilloma excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pterygium operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days